CLINICAL TRIAL: NCT04194879
Title: Effectiveness of Multi-target FIT-DNA Analysis as a Colorectal Cancer Screening Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Dominic C.C. Foo, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 19-784
Record Dates: First submitted 2019-12-08; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer; Adenoma Colon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer: Case subjects (at least 50) will be men and women age 40-74 who are recently diagnosed, through colonoscopy, with different stages of colorectal cancer and have not yet had surgical intervention.
  Interventions: Diagnostic Test: multi-target FIT-DNA analysis
- Negative: Approximately 250 prospectively enrolled subjects will be men and women age 40-74 who are at average risk of developing colorectal cancer and eligible for colonoscopy. About 150 Control subjects will be enrolled prospectively, who have no colorectal neoplasia detected on colonoscopy, including cancer, advanced adenoma, sessile serrated lesions and small, non-advanced adenoma.
  Interventions: Diagnostic Test: multi-target FIT-DNA analysis

INTERVENTIONS:
Diagnostic Test: multi-target FIT-DNA analysis — ColoClear® is intended for use as an adjunctive screening test for the detection of colorectal neoplasia associated DNA markers and for the presence of occult hemoglobin in human stool. It has the potential of increasing the sensitivity of detecting CRC as compared to FOBT or faecal immunochemical test (FIT), which detects the presence of hemoglobin in stool alone. A positive result may indicate the presence of colorectal cancer or pre-malignant colorectal neoplasia. ColoClear® is not intended as a replacement for diagnostic colonoscopy. A positive result in ColoClear®, as with any screening test, should be followed by colonoscopy. ColoClear® is intended for colorectal cancer screening in average risk individuals: adults of either sex, 40 years or older, who are at high risk for colorectal cancer.
  Other Names: Coloclear

SUMMARY:
Colorectal cancer is one of the most common cancer in Hong Kong. In 2018, CRC accounted for 17.4%, 5,780 cases, of the total new cancers. CRC claimed 2,279 lives (15.8%) making it the second most deadly killer in the population.

Since 2010, the Cancer Expert Working Group (CEWG) has recommended that asymptomatic average-risk individuals aged 50 to 75 years should consider one of the screening methods: fecal occult blood test (FOBT) every one to two years; OR flexible sigmoidoscopy every 5 years; OR colonoscopy every 10 years. However, it poses great challenges for large scale CRC screening using colonoscopy, such as bowel preparation difficulties, complications of procedure and poor compliance.

ColoClear® is intended for use as an adjunctive screening test for the detection of colorectal neoplasia associated DNA markers and for the presence of occult hemoglobin in human stool. It has the potential of increasing the sensitivity of detecting CRC as compared to FOBT or faecal immunochemical test (FIT), which detects the presence of hemoglobin in stool alone. A positive result may indicate the presence of colorectal cancer or pre-malignant colorectal neoplasia. ColoClear® is not intended as a replacement for diagnostic colonoscopy. A positive result in ColoClear®, as with any screening test, should be followed by colonoscopy. ColoClear® is intended for colorectal cancer screening in average risk individuals: adults of either sex, 40 years or older, who are at high risk for colorectal cancer.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the clinical performance of ColoClear test in early screening of colorectal cancer in Hong Kong. Other outcomes to analyze include, but are not limited to the point estimate of the sensitivity of ColoClear for the detection of advanced adenoma (AA) in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at average risk for development of CRC.
* Subject is male or female (all Asian), 40-74 years of age.
* Subject is able to comprehend, sign and date the written informed consent form to participate in this study, undergo study procedures described in the informed consent form and authorizes release of relevant protected health information through signing an informed consent form.

Exclusion Criteria:

* Subject undergone colonoscopy and removal of lesions within 5 years.
* Subject with Familial Adenomatous Polyposis (FAP) and Inflammatory Bowel Disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease.
* Subject with overt rectal bleeding, e.g., hematochezia or melena, within the previous 30 days.
* Any condition which, in the opinion of the investigator should preclude participation in the study.

Ages: 40 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 300 subjects (assume 20% drop out rate)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity & specificity of colorectal cancer detection | within 3 months
  The primary endpoint is the point estimate of sensitivity and specificity of ColoClear for screening of CRC.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic CC Foo, MBBS, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The data could be stored in a public repository for other researchers after completion